CLINICAL TRIAL: NCT02508831
Title: Double Upper Limb Allograft: Intervention and Clinical Evaluation. A Pilot Study of 5 Cases
Acronym: DAMIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL14_0199
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Bilateral Amputation of Upper Limb
Keywords: Bilateral amputation; upper limb; allograft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bilateral amputation of upper limb (Experimental): Patients with bilateral amputation of upper limb will receive a double upper limb allograft
  Interventions: Procedure: Double upper limb allograft

INTERVENTIONS:
Procedure: Double upper limb allograft — Patients with bilateral amputation of upper limb will receive a double upper limb allograft

SUMMARY:
The case of patients with amputation of forearm on one side and arm on the other is particularly interesting to study because in this situation of handicap greater than a double amputation in forearm. We should bring a functional benefit to the patient with the transplant of forearm and this situation allows to have the best possible control to compare the result of the transplant of arm to that of forearm because it is realized at the same patient.

Amputation of both arms deprives patients of an elbow what establishes a major factor of limitation of autonomy and makes patients totally dependent for the realization of the essential gestures of the current life requiring the prehension (dress, dressing, food, hygiene of the elimination). The various equipments are not always adaptable and usable. Psychologically, an amputation in arm is unanimously considered as an infringement very badly accepted of the physical integrity and establishes a major handicap factor of family, professional and social exclusion.

The results of this study should allow a better appreciation of indications and modalities of care of biamputed patients with at least one lesion level above the elbow.

This clinical research will determine the potential place of a reconstructive surgery as allograft in biamputed patients on the basis of functional results and assessment of disorders of the body schema perception.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Bilateral amputation of upper limb regardless of the nature of the injury (crush, tearing, cutting, infectious such as purpura fulminans...) except for tumor diseases
* Lesion level:

  * The non-transplant patients-free immunosuppressive therapy: bilateral amputation of upper limb with at least one lesion level above the elbow. Higher amputation level is fixed to the upper 1/4 of the arm to allow for a recovery of active flexion of the elbow against gravity.
  * For organ transplant patients (other than hand or upper extremity: ex liver, kidney) and already under bi - or tri-therapy immunosuppressive : bilateral amputation of upper limb with at least one lesion level above the elbow. The top level of amputation may be above the upper 1/4 of the arm especially if body image disorders dominate the complaint of the patient.
* Period since amputation of at least 6 months
* Failure of all currently available (including the prosthetic) support modalities
* Psychological maturity: absence of serious disorder of the personality or chronic disorders of mood reported by psychiatrists of the team using tests for the assessment of personality, committed and voluntary patients
* Signature of the free and informed consent form

Exclusion Criteria:

* Mono-amputee patient
* Patients with brachial plexus lesions
* Patients with vascular disorders likely result in thrombosis
* Active smoking patients
* Patients in an emergency medical situation
* Antecedent of malignant tumor in remission for less than 5 years
* Patients with malignant tumor
* Patients with a American Society of Anesthesiology (ASA) score > 3
* Patients with glomerular filtration < 60 ml/min
* Patients with severe hypertension : Systolic Blood Pressure (SBP) > 140 mmHg and Diastolic Blood Pressure (DBP) > 90 mmHg

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2016-07-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Changes in functional recovery from baseline to 5 years after the transplant of upper limbs | Before the transplant, then at 6 months, 1, 2, 3, 4 and 5 years after a double transplant of upper limbs.
  Functional results assessed by a multidimensional evaluation:
  * A general clinical assessment
  * An analytical assessment:
    * Articular : Total Active Motion (TAM) as a percentage of Total Passive Motion (TPM)
    * Muscle: manual muscle strength testing and quantitative by Jamar dynamometers
  * A sensory and proprioceptive balance: sensitivity on mapping of WINN-PARRY, with assessment of sensitivity of protection and discriminative touch mobile and static touch, Moving Two Points Distance, Static Two Points Distance (Weber test).
  * A functional balance based on: DASH test, Carroll test, balance of 400 points, tests of independence and Hand Transplantation Score System (HTSS)
  * Impact on quality of life: measured by the Medical Outcome Study Short Form-36 (MOS SF-36)

SECONDARY OUTCOMES:
Patients body image perception | To be measured before the transplant, then at 6 months, 1, 2, 3, 4 and 5 years after transplant
  An auto-questionnaire based on 3 questions answered by level type Likert (not at all agree, disagree, neutral, agree, quite agree)
  • Questionnaire Fragebogen zum KorperBild 20 (FKB-20)
Patients' self-esteem | To be measured before the transplant, then at 6 months, 1, 2, 3, 4 and 5 years after transplant
  The Rosenberg self-esteem scale will be used to evaluate patients amputated and then grafted.
Brain plasticity post-transplant | Before intervention, then 3, 6, 12, 18 and 24 months after the transplant.
  The degree of reorganization of the primary motor cortex will be measured by the assessment of re-innervation and the integration of the graft to the body schema by cerebral functional MRI with psychological tests.
Acute rejection rate in post-transplant period | To be measured at 6 months, 1, 2, 3, 4 and 5 years after transplant
  To be appreciated by inflammatory signs (erythema) at the clinical examination. The diagnosis of acute rejection will be confirmed on the basis of histological results.
Chronic rejection rate in post-transplant period | Throughout the five years of follow-up
  To be approached by various exams:
  * MRI
  * CT scan of segments transplanted
  * Micro-Doppler looking for intimal hypertrophy
  * An endovascular echography of vessels above the fold of the elbow
  * Capillaroscopy
  * Arteriography will be carried out at 5 years to better appreciate achieving vascular grafts
  * Histological study of the skin and deep tissues.
Walking analysis in posturography | To be carried out before the transplant, then at 6 months, 1, 2, 3, 4 and 5 years after transplant
  The walking analysis is a non-invasive examination which consist in recording the movements by a roptoelectronic device. This system captures the three-dimensional position of retro-reflective markers placed on the body. Once analyzed, this information allows getting data quantified on movements.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - Service d'Urologie et Chirurgie de la Transplantation, Lyon, France